CLINICAL TRIAL: NCT05098951
Title: Efficacy and Safety of Acupuncture for Relieving Stiffness of Joint Related to Aromatase Inhibitors in Patients With Early-Stage Breast Cancer
Brief Title: Acupuncture for Stiffness of Joint Related to Aromatase Inhibitors in Patients With Early-Stage Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AHQU-2021004
Record Dates: First submitted 2021-10-17; First posted 2021-10-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Stiffness of Hand, Not Elsewhere Classified
Keywords: Breast cancer; Stiffness; Aromatase inhibitor; Acupuncture; High altitude
MeSH Terms: conditions — Breast Neoplasms; Altitude Sickness | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with stiffness of joint receive acupuncture therapy (Experimental): This is a single arm study. All the enrolled patients will receive acupuncture twice weekly for 6 weeks then once weekly for another 6 weeks.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Patients with stiffness of joint receive acupuncture therapy twice weekly for 6 weeks and then once weekly for 6 weeks.

SUMMARY:
RATIONALE: Acupuncture may help relieve joint stiffness related to aromatase inhibitors in patients with early-stage breast cancer.

PURPOSE: This single arm clinical study aims to evaluate how well acupuncture as a non-pharmacological treatment, works in treating patients with joint stiffness related to aromatase inhibitors (AIs) in patients with early-stage breast cancer.

DETAILED DESCRIPTION:
Objectives of this study:

Primary objective:

To evaluate whether acupuncture as a non-pharmacological treatment, administered twice weekly for 6 weeks can significantly reduce joint stiffness related to AIs in women with early-stage breast cancer as measured by the Western Ontario and McMasters Universities Osteoarthritis (WOMAC) stiffness score at weeks 6.

Secondary objectives:

To evaluate the effect of acupuncture on joint stiffness measured by the WOMAC stiffness score at weeks 12.

To evaluate the effect of acupuncture on joint stiffness measured by the Modified Score for the Assessment of Chronic Rheumatoid Affections of the Hands (M-SACRAH) stiffness score at weeks 6 and weeks 12.

To evaluate the effects of acupuncture on quality of life (QOL) assessed by the Functional Assessment of Cancer Therapy-Endocrine Subscales (FACT-ES) at weeks 6 and weeks 12.

To evaluate the safety and tolerability of acupuncture in the enrolled patients.

To identify potential genetic determinants to response to acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. History of stage I-III breast cancer and free of disease by clinical examination
2. Postmenopausal or premenopausal with ovarian suppression
3. Currently receiving aromatase inhibitors (Anastrozole, Letrozole, or Exemestane) treatment
4. With joint stiffness attributed to the use of aromatase inhibitors
5. Having had joint stiffness for at least 1 months
6. Having had at least 15 days with stiffness in the preceding 30 days

Exclusion Criteria:

1. Women with recurrent or metastatic breast cancer
2. Women having finished chemotherapy or radiation therapy less than 1 months prior to enrollment
3. Women with history of bleeding disorder
4. Women with joint stiffness attributed to inflammatory arthritis, such as rheumatoid arthritis, spondy loarthritis and osteoarthritis
5. Women having joint stiffness prior to AI treatment
6. Women that have received treatment of any kind for joint stiffness within the last 3 months
7. Women that have previously received the acupuncture treatment before for any reason

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study just enroll female patients with breast cancer.
Enrollment: 52 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The change in stiffness score as measured by the Western Ontario and McMasters Universities Osteoarthritis (WOMAC) | 6 weeks
  The change in stiffness score as measured by the Western Ontario and McMasters Universities Osteoarthritis (WOMAC) at the end of week 6 of intervention compared to that at baseline.

SECONDARY OUTCOMES:
The change in stiffness score as measured by the Modified Score for the Assessment of Chronic Rheumatoid Affections of the Hands (M-SACRAH) | 6 weeks
  The change in stiffness score as measured by the Modified Score for the Assessment of Chronic Rheumatoid Affections of the Hands (M-SACRAH) at the end of week 6 of intervention compared to that at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jiuda Zhao, Principal Investigator — the Affiliated Hospital of Qinghai University
Locations (1):
- Affiliated Hospital of Qinghai University, Affiliated Cancer Hospital of Qinghai University, Xining, Qinghai, China